CLINICAL TRIAL: NCT05768841
Title: Prevalence of Mental Health Issues in Endurance Athletes.
Status: Recruiting | Type: Observational
Sponsor: Ultra Sports Science Foundation (Other)
Collaborators: Hospital Universitario del Vinalopo (Unknown); Universidade do Porto (Other); University of South Africa (Other)
Responsible Party: Principal Investigator, Volker Scheer, Professor, Ultra Sports Science Foundation
Other Study IDs: VS1
Record Dates: First submitted 2023-03-03; First posted 2023-03-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Depression, Anxiety; Mental Health Issue
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- endurance athletes: participants that have or are participating in endurance sports
  Interventions: Behavioral: mental health issues

INTERVENTIONS:
Behavioral: mental health issues — survey on mental health issues in endurance athletes

SUMMARY:
Participation in endurance sports has been increasing over the last few decades and our aim of our exploratory descriptive survey study is therefore to examine mental health issues in endurance athletes (marathon runners, ultra endurance runners, triathletes), employing the IOC assessment tool, to provide information on mental health issues in this population. Secondary objects are to evaluate risk factors for mental health issues in endurance athletes (like exercise behaviour, competition behaviour, age, gender, medical issues)

DETAILED DESCRIPTION:
This study is an exploratory descriptive survey study.

The study protocol will be largely replicated from the IOC consensus paper and the questionnaires based according to SMHAT 1 with an athlete-specific screening tool (APSQ) and further eleven subsequent disorder-specific screening tools:

Eleven disorder specific screening tools:

1. General Anxiety Disorder-7 (GAD-7): assesses the presence of symptoms of anxiety.
2. Patient Health Questionnaire-9 (PHQ-9): assesses the presence of symptoms of depression.
3. Athlete Sleep Screening Questionnaire (ASSQ): assesses the presence of sleep disturbance.
4. Alcohol Use Disorders Identification Test Consumption (AUDIT-C): assesses the presence of alcohol misuse.
5. Cutting Down, Annoyance by Criticism, Guilty Feeling, and Eye-openers Adapted to Include Drugs (CAGE-AID): assesses the presence of substance misuse, being slightly adapted for the SMHAT (no focus on alcohol use as already explored with the AUDIT-C; additional question to explore which substance was used).
6. Brief Eating Disorder in Athletes Questionnaire (BEDA-Q): assesses the presence of disordered eating.
7. ADHD
8. Bipolar disorder
9. PTSD
10. Gambling
11. Psychosis

Additionally questions to assess exercise addiction will be used as it has been shown that exercise addiction may be particularly prevalent in endurance athletes.

Further questions about age, gender, country of origin, training data, past medical history and medication will be asked as well as a few specific questions about there thoughts on mental health issues as per IOC consensus paper

ELIGIBILITY:
Inclusion Criteria:

* endurance athletes (marathon runners, ultramarathon runners and triathletes)
* over the age of 16
* all genders
* recreational athletes (non- elite)
* elite athletes (professional, international, college level)

Exclusion Criteria:

* athletes that that are not competing or have not competed in an official endurance race
* athletes that are younger than 16 years of age.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Particpants that have or are participating in endurance sports
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with mental health issues | March-September 2023
  Number of participants with mental health issues

SECONDARY OUTCOMES:
Number of participants with risk factors associated with mental health issues | March-September 2023
  Number of participants with risk factors associated with mental health issues

CONTACTS AND LOCATIONS:
Overall Officials: Volker Scheer, Prof, Principal Investigator — Ultra Sports Science Foundation
Locations (1):
- Ultra Sports Science Foundation, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No
anonymous